CLINICAL TRIAL: NCT01318837
Title: Reproducibility Study of OABSS and Its Response to Solifenacin Treatment (RESORT) and Validity in Korean Populations; Part 2: Responsiveness and Validity
Brief Title: A Study to Evaluate Response of Over Active Bladder Symptom Score to Solifenacin Treatment
Acronym: RESORT-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: OABSSVSK-002
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Over Active Bladder
Keywords: OABSS; IPSS; PPBC; Solifenacin
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sofilenacin group (Experimental)
  Interventions: Drug: solifenacin
- control group (No Intervention): age and sex matched patients without OAB symptom who will answer demographic questionaire and OABSS once

INTERVENTIONS:
Drug: solifenacin — oral
  Other Names: Vesicare
  Arms: sofilenacin group

SUMMARY:
This study is to evaluate change of over active bladder symptom scores (OABSS) between, before and after solifenacin treatment to OAB subjects.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB for 3 months or longer
* At least 1 urgency episode in last 3 days
* Symptoms of OAB as verified by the screening 3-day bladder diary, defined by:

  * a. Number of micturition ≥8 times/day
  * b. Number of urgency episodes in 3 days ≥3

Exclusion Criteria:

* Significant stress incontinence or mixed stress/urge incontinence
* Subject with indwelling catheters or practicing intermittent self-catheterization
* Symptomatic urinary tract infection, chronic inflammation
* Diabetic neuropathy
* Subjects who are prohibited from taking solifenacin as contraindications
* Drug or non-drug treatment for OAB was started, quitted or changed in 4 weeks
* Participation in any clinical trial in 30 days except for Part-1 of RESORT
* Diabetic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to week 4 in Over-Active Bladder Symptom Score (OABSS) | week 0 (baseline) and week 4
Changes from baseline to week 12 in OABSS | week 0 (baseline) and week 12

SECONDARY OUTCOMES:
Changes from baseline in International Prostate Symptom Score (IPSS) at week 4 | week 0 (baseline) and week 4
Changes from baseline in IPSS at week 12 | week 0 (baseline) and week 12
Changes from baseline in Quality of Life (QoL) Score at week 4 | week 0 (baseline) and week 4
Changes from baseline in QoL Score at week 12 | week 0 (baseline) and week 12
Changes from baseline in Patient Perception of Bladder Condition (PPBC) at week 4 | week 0 (baseline) and week 4
Changes from baseline in PPBC at week 12 | week 0 (baseline) and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Principal Investigator — Bundang Seoul National University Hospital, Seong Jin Jeong, MD.
Locations (2):
- South Korea (2):
  - Seoul
  - Sungnam

REFERENCES:
- [Background] Jeong SJ, Homma Y, Oh SJ. Reproducibility study of Overactive Bladder Symptom Score questionnaire and its response to treatment (RESORT) in Korean population with overactive bladder symptoms. Qual Life Res. 2014 Feb;23(1):285-92. doi: 10.1007/s11136-013-0440-7. Epub 2013 May 29. PMID 23715806